CLINICAL TRIAL: NCT04779775
Title: Best Practices in Perinatal Mental Health During COVID-19 Pandemic: A Collaborative Research Study Between the COST Actions RISEUP-PPD and Devotion
Brief Title: Best Practices in Perinatal Mental Health During COVID-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Minho (Other)
Collaborators: Universidad Loyola Andalucia (Other); Catholic University of Croatia (Unknown); University of Coimbra (Other)
Responsible Party: Principal Investigator, Ana Mesquita, Principal Investigator, University of Minho
Other Study IDs: RISEUP-PPD-DEVOTION- COVID-19
Record Dates: First submitted 2021-02-10; First posted 2021-03-03 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Perinatal Mental Health Care Practices During the COVID-19 Pandemic
Keywords: perinatal mental health policies; guidelines; protocols; perinatal care practices; best practices during COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The COVID-19 pandemic has caused changes in health care during pregnancy, childbirth and postpartum. Although adverse effects of COVID-19 on perinatal mental health have been documented, changes in the perinatal mental health care provided to women and their families are yet to be established. As a Task Force in Perinatal mental health and COVID-19 pandemic within RISEUP-PPD COST Action, we aim: (i) to identify policies, guidelines and protocols from different European countries concerning the provision of perinatal mental health care in face of COVID-19, and (ii) to select the best practices to alleviate the negative impact of COVID-19 on perinatal mental health. The survey will be conducted among experts in perinatal mental health who are members of the COST Action RISEUP-PPD and COST Action Devotion in 36 European countries. The experts will fill in the online survey designed for this study that includes a series of open-ended questions, checklists, and response ratings on a 7-point scale. The topic areas cover seven domains of interest: 1) mental health policies, guidelines, protocols, and documents; 2) mental health care practices; 3) best practices; 4) barriers; 5) resources; 6) benefits; and 7) short- and long-term expectations. Data analysis will be mainly a qualitative analysis of the experts' professional views and opinions about the policies, guidelines, protocols, and documents regarding perinatal mental health changes in their country. Additionally, a basic quantitative descriptive analysis will be conducted.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is an infectious disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) that has caused worldwide pandemic since the breakout from Wuhan, China in December 2019. It has infected more than 71.5 million people, causing 1.6 million of deaths up to mid of December 2020.

Perinatal health care practices have been changed for safety reasons due to the pandemic and are still changing locally according to the epidemiological circumstances. Across Europe antenatal classes have ceased or have been provided online, antenatal regular check-ups are somewhat reduced or offered via telephone, the presence of the supporting person during childbirth is often not allowed in a maternity ward, visits of the father and other family members to the hospital after delivery are reduced or restricted, newborns of infected mothers are sometimes separated, home visits of a midwife after birth and breastfeeding support are also reduced (COST Devotion). Although official and national guidelines for perinatal health in general or infected mothers/newborns may be available, practices have been changing constantly, some of which may not be evidence-based or are in contradiction with the recommendations. Along with these changes, there are general restrictions, such as distancing from others, restricted socializing, and restricted movement, which may be necessary but can impose substantial psychological distress.

The high impact of COVID-19 on maternal mental health during pregnancy and postpartum has been evident in different countries worldwide. All these changes due to COVID-19 pandemic and related epidemiological measures were necessary to combat the spread of the virus but lead to an adverse effect on perinatal mental health.

Within the ongoing COST Action Research Innovation and Sustainable Pan-European Network in Peripartum Depression Disorder - RISEUP-PPD, funded by the European Cooperation in Science and Technology (COST Association), the special Task Force Perinatal mental health and COVID-19 pandemic, in collaboration with the COST Action Perinatal Mental Health and Birth-Related Trauma: Maximising best practice and optimal outcomes - Devotion, has been established with the main aim of investigating the best practices and guidelines to alleviate the negative consequences of COVID-19 on women's mental health (RISEUP-PPD COST Action). A recent review pointed out emerging issues in the prevention, diagnosis, and treatment of peripartum depression, which are highlighted even more with the ongoing pandemic. The Task Force has already addressed the deleterious impact of COVID-19 on perinatal mental health, the risk factors for mental health vulnerability during the current pandemic and highlighted good psychological practices in perinatal mental health during the COVID-19 pandemic. The Task Force pointed out that research on good practices in perinatal mental health in the time of COVID-19 pandemic should (i) capture the wide range of psychological distress presentations, focusing on depression and anxiety, (ii) look into complex roles of physical distancing and social isolation due to epidemiological measures, (iii) take into account the barriers in seeking help augmented by the pandemic that may be overcome by new e-health services, (iv) investigate changes in perinatal healthcare practices and factors that may alleviate them, and finally (v) boost the efforts for further development and validation of specific perinatal mental health assessment tools.

However, it remains yet to investigate what are the good practices in perinatal mental health and how have those been incorporated in the national policies, guidelines, protocols, and official documents across European countries during the COVID-19 pandemic. This has important clinical implications and can be used to inform policymakers at both the national and the European level - with the ultimate goal of providing the adequate support to women in the peripartum period and promote a pleasant experience for mothers and their families during pregnancy, delivery and the postpartum, in particular challenging situations as it is the case of the present COVID-19 pandemic. The main aim of this study is to identify the best practices to alleviate the negative impact of COVID-19 itself and the related safety measures (in health care facilities) and to promote mental health support during perinatal period. The secondary aim is to identify the themes emerging from the experts' opinions on changes due to COVID-19 pandemic in 1) mental health policies, guidelines, protocols, and documents; 2) mental health care practices; 3) best practices; 4) barriers; 5) resources; 6) benefits; and 7) short- and long-term expectations.

Methods and analysis Study design A cross- sectional study will be conducted in order to identify best practices in perinatal mental health during the COVID-19 pandemic.

Participants The participants will be experts in perinatal mental health who are the members of the COST Action RISEUP-PPD and the COST Action Devotion. The COST members are applied sciences researchers and clinicians (nurses, midwives, clinical social workers, general practitioners, Obstetrician/Gynaecologist, psychiatrists, clinical psychologist, psychotherapists), added by researchers from other backgrounds such as neuroscience, biology, biomedical engineer, mathematics and statistics, etc.), politicians, decision-makers, peer-support groups, stakeholders. The main aim of the RISEUP-PPD is to gather a multidisciplinary network of researchers to collect and profound the knowledge about prevention, assessment, and treatment in peripartum depression, while Devotion is dedicated to minimising birth trauma and optimising birth experiences. Taken together, both COST Actions include representatives from 35 European COST countries (Albania, Austria, Belgium, Bosnia and Herzegovina, Bulgaria, Croatia, Cyprus, Czech Republic, Denmark, Estonia, Finland, France, Germany, Greece, Iceland, Ireland, Italy, Latvia, Lithuania, Luxembourg, Malta, Netherlands, North Macedonia, Norway, Poland, Portugal, Romania, Serbia, Slovakia, Slovenia, Spain, Sweden, Switzerland, Turkey, United Kingdom), Israel as a Cooperating Members, and Brazil, the USA, Canada and Australia as International Partner countries.

As mainly qualitative data is planned to be collected, no calculation on sample size is necessary.

Instruments Demographic and expertise background questionnaire The Demographic and expertise background questionnaire will comprise questions on the area of specialisation (Nurse, Midwife, Clinical social worker, General practitioner, Obstetrician/Gynaecologist, Psychiatrist, Psychologist, Psychotherapist, Other), academic background and degree, job position in the current institution, years of experience and years working in Perinatal Care and/or Perinatal Mental Health (each with categories: up to 1 year, 2-5 years, 5-10 years, more than 10 years), current employer (tick all that apply: public, private, birth centre, hospital, home birth, primary care service, academic/research, counselling office, non-governmental organization, other), number of patients/clients per year per institution and personally, gender, age and country.

Questionnaire for experts on perinatal mental health practices during the COVID-19 Pandemic A questionnaire for the consultation of experts was developed by the research group of the Task Force "Perinatal Mental Health and COVID-19 pandemic", based on the previous questionnaire for experts on mental health used in Europe. The questionnaire includes a series of open-ended questions, checklists, and response ratings on a 7-point scale (1 = not adequate to 7 = excellent) with specific references to the change of policies, protocols, and practices regarding Perinatal Mental Health during COVID-19 pandemic. The topic areas covered seven domains of interest: 1) mental health policies, guidelines, protocols, and documents; 2) mental health care practices; 3) best practices; 4) barriers; 5) resources; 6) benefits; and 7) short- and long-term expectations.

Guidelines are defined as systematically developed recommendations to assist in practitioner and patient decision making about treatments for clinical conditions. Protocols are a comprehensive set of criteria outlining the management steps for a single clinical condition. Documents are defined as official records that provide information or evidence. Finally, Best Practice is defined as a technique or methodology that through experience and research has proven reliably to lead to the desired result.

The survey was written in English and a pilot study with three experts in perinatal mental health was conducted. Questions for pilot are presented in Table in Appendix 1. Amendments to the questionnaire were made accordingly which included rewording questions to elicit appropriate responses. The questionnaire for key experts can be found in Appendix 2.

Procedure Experts from COST Action RISEUP-PPD and COST Action Devotion will be approached by e-mail invitation to participate in the study. In order to have greater representation, the research group will encourage that, at least, the three experts per country with more expertise received the invitation.

Experts will be asked to complete the questionnaire online (Qualtrics platform). First, they will read an electronic consent form presenting an overview of the study aims, content of the questions asked, potential risks and benefits, and ethical aspects of the study (i.e., voluntary participation, confidentiality and secure storage of the data, and absence of any type of compensation). At the bottom of the form, they will be asked to confirm a eligibility criteria (members of either COST Actions) and to provide their consent to participate in the study. Participants who do not meet the predefined inclusion criteria will be directed to a message thanking them for their interest and informing them of the required eligibility criteria for participation in the study. The questionnaires are estimated to take approximately 15-20 minutes to complete.

Data analysis Data analysis will be mainly a qualitative analysis of the experts' views and opinions about the policies, guidelines, protocols, and documents regarding perinatal mental health changes in their country. The analysis will be made across the seven dimensions: 1) mental health policies, guidelines, protocols, and documents; 2) care practices; 3) best practices; 4) barriers; 5) resources; 6) benefits; and 7) short- and long-term expectations. Two authors will develop the coding plan, which will be checked by other authors. Two authors will code all answers to the open-ended questions independently. Inter-rater reliability will be calculated by Cohen's kappa coefficient and all disparities will be discussed to the agreement.

Additionally, a basic quantitative descriptive analysis will be made to estimate how many experts think that the policies, guidelines, or protocols regarding perinatal mental health have changed since COVID-19 outbreak, including percentages of yes/no answers and central tendency/variance on 7-point scale answers.

The findings from this study will be disseminated as papers published in peer-reviewed journals, presented at national and international conferences, and most importantly, its results will be used inform policymakers and have an impact on the changes in perinatal mental health care on a national and European level.

ELIGIBILITY:
Inclusion Criteria:

* experts working in perinatal care services within the COST actions RISEUP-PPD and Devotion

Exclusion Criteria:

* COST members working in perinatal mental health less than 1 year

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Experts in perinatal mental health who are the members of the COST Action RISEUP-PPD and the COST Action Devotion
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in perinatal best practices | March 2020- June 2021
  Questionnaire on changes in perinatal mental health care practices during the COVID-19 Pandemic
Changes in perinatal mental health protocols | March 2020- June 2021
  Questionnaire on changes in perinatal mental health care practices during the COVID-19 Pandemic

CONTACTS AND LOCATIONS:
Overall Officials: Ana Mesquita, PhD, Principal Investigator — University of Minho; Emma Motrico, PhD, Principal Investigator — University of Loyola; Sandra Nakić Radoš, PhD, Principal Investigator — Catholic University of Croatia; Ana Ganho, PhD, Principal Investigator — University of Coimbra; Joan Lalor, PhD, Principal Investigator — Trinity College of Dublin

REFERENCES:
- [Background] Brooks SK, Webster RK, Smith LE, Woodland L, Wessely S, Greenberg N, Rubin GJ. The psychological impact of quarantine and how to reduce it: rapid review of the evidence. Lancet. 2020 Mar 14;395(10227):912-920. doi: 10.1016/S0140-6736(20)30460-8. Epub 2020 Feb 26. PMID 32112714
- [Background] Chen D, Yang H, Cao Y, Cheng W, Duan T, Fan C, Fan S, Feng L, Gao Y, He F, He J, Hu Y, Jiang Y, Li Y, Li J, Li X, Li X, Lin K, Liu C, Liu J, Liu X, Pan X, Pang Q, Pu M, Qi H, Shi C, Sun Y, Sun J, Wang X, Wang Y, Wang Z, Wang Z, Wang C, Wu S, Xin H, Yan J, Zhao Y, Zheng J, Zhou Y, Zou L, Zeng Y, Zhang Y, Guan X. Expert consensus for managing pregnant women and neonates born to mothers with suspected or confirmed novel coronavirus (COVID-19) infection. Int J Gynaecol Obstet. 2020 May;149(2):130-136. doi: 10.1002/ijgo.13146. Epub 2020 Apr 1. PMID 32196655
- [Background] Ciotti M, Ciccozzi M, Terrinoni A, Jiang WC, Wang CB, Bernardini S. The COVID-19 pandemic. Crit Rev Clin Lab Sci. 2020 Sep;57(6):365-388. doi: 10.1080/10408363.2020.1783198. Epub 2020 Jul 9. PMID 32645276
- [Background] COST Action "Devotion": Perinatal Mental Health and Birth Related Trauma: Maximising Best Practices and Optimal Outcomes. (2020). COVID in different countries - group discussion.
- [Background] Davenport MH, Meyer S, Meah VL, Strynadka MC, Khurana R. Moms Are Not OK: COVID-19 and Maternal Mental Health. Front Glob Womens Health. 2020 Jun 19;1:1. doi: 10.3389/fgwh.2020.00001. eCollection 2020. PMID 34816146
- [Background] European Commission. (2013). Mental health systems in the European Union member states, status of mental health in populations and benefits to be expected from investments into mental health main report. (July), 1-574.
- [Background] Fonseca A, Ganho-Avila A, Lambregtse-van den Berg M, Lupattelli A, Rodriguez-Munoz MF, Ferreira P, Rados SN, Bina R. Emerging issues and questions on peripartum depression prevention, diagnosis and treatment: a consensus report from the cost action riseup-PPD. J Affect Disord. 2020 Sep 1;274:167-173. doi: 10.1016/j.jad.2020.05.112. Epub 2020 May 23. PMID 32469800
- [Background] Motrico, E., Mateus, V., Bina, R., Felice, E., Bramante, A., Kalcev, G., ... & Mesquita, A. Good practices in perinatal mental health during the COVID-19 pandemic: a report from Task-force RISEUP-PPD COVID-19. Clínica y Salud. 2020; 31(3), 155-160.
- [Background] Queensland Clinical Guidelines (2020). Perinatal care of suspected or confirmed COVID-19 pregnant women. Guideline No. MN20.63-V2-R25. Queensland Health. Available from: http://www.health.qld.gov.au/qcg
- [Background] Saccone G, Florio A, Aiello F, Venturella R, De Angelis MC, Locci M, Bifulco G, Zullo F, Di Spiezio Sardo A. Psychological impact of coronavirus disease 2019 in pregnant women. Am J Obstet Gynecol. 2020 Aug;223(2):293-295. doi: 10.1016/j.ajog.2020.05.003. Epub 2020 May 7. No abstract available. PMID 32387321
- [Background] Thapa SB, Mainali A, Schwank SE, Acharya G. Maternal mental health in the time of the COVID-19 pandemic. Acta Obstet Gynecol Scand. 2020 Jul;99(7):817-818. doi: 10.1111/aogs.13894. No abstract available. PMID 32374420
- [Background] Topalidou A, Thomson G, Downe S. COVID-19 and maternal mental health: Are we getting the balance right? medRxiv. 2020; https://doi.org/10.1101/2020.03.30.20047969
- [Background] World Health Organization [WHO] (2020a). WHO Coronavirus Disease (COVID-19) Dashboard. https://covid19.who.int/ Accessed 16 December 2020.
- [Background] Thomson S, Doan T, Liu D, Schubert KO, Toh J, Boyd MA, Galletly C. Supporting the vulnerable: developing a strategic community mental health response to the COVID-19 pandemic. Australas Psychiatry. 2020 Oct;28(5):492-499. doi: 10.1177/1039856220944701. Epub 2020 Jul 30. PMID 32729320
- [Derived] Rados SN, Motrico E, Mesquita AM, Ganho-Avila A, Vousoura E, Lalor J. Changes in perinatal mental healthcare during the COVID-19 pandemic: a protocol for a collaborative research study between the COST actions RISEUP-PPD and DEVOTION. BMJ Open. 2022 Jul 26;12(7):e052411. doi: 10.1136/bmjopen-2021-052411. PMID 35882459